CLINICAL TRIAL: NCT05305352
Title: Very Low Carbohydrate Dietary Intervention in Gestational Diabetes Mellitus: Effect on Glycemic, Metabolic, Glycated and Inflammatory Marker: A Randomized Controlled Trial
Brief Title: Effect of Very Low Carbohydrate Diet on Glycemic, Metabolic, Glycated and Inflammatory Markers in Gestational Diabetes Mellitus
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to less number of participants willing to participate.
Sponsor: Khyber Medical University Peshawar (Other)
Responsible Party: Principal Investigator, Bibi Hajira, Assistant Professor, Khyber Medical University Peshawar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DIR/KMU-AS&RB/EV/001551
Record Dates: First submitted 2022-02-28; First posted 2022-03-31 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Gestational Diabetes; Inflammation; Metabolic Syndrome; Glucose Intolerance During Pregnancy; Glucose Intolerance; Insulin Resistance
Keywords: gestational diabetes; insulin resistance; carbohydrate; inflammation; glucose intolerance
MeSH Terms: conditions — Diabetes, Gestational; Inflammation; Metabolic Syndrome; Glucose Intolerance; Insulin Resistance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No intervention (No Intervention): The no intervention arm will not receive counselling but will follow their routine diet suggested during their routine antenatal visits.
- Intervention (Experimental): The intervention arm will be counselled about very low carbohydrate diet (<10%carbohydrate)
  Interventions: Other: Very low carbohydrate dietary intervention

INTERVENTIONS:
Other: Very low carbohydrate dietary intervention — The experimental group will be counseled about very low carbohydrate diet i.e., <10% carbohydrate,40-50% protein and lipid in diet).
  Arms: Intervention

SUMMARY:
Uncontrolled Gestational Diabetes Mellitus may leads to maternal and fetal complications. These complications can be avoided by adopting the dietary modifications along with medications. Previous studies suggested that consumption of low Carbohydrate diet improves Gestational Diabetes and related complications. Therefore, this study aims to investigate the effect of very low carbohydrate dietary intervention on glycemic, glycemic, metabolic, glycated and inflammatory markers.

DETAILED DESCRIPTION:
This will be randomized controlled trial of 80-100 Gestational diabetic women of second trimester to investigate the effect of very low carbohydrate dietary intervention on glycemic, metabolic, glycated and inflammatory markers.

Subjects will be recruited from ob/gyn outpatient of different hospitals. Eligible subjects will be enrolled in the study and will be allocated into two groups. One will be intervention and other will be control group. At baseline fasting blood samples from both group will be taken and will be analyzed for different biomarkers. Thereafter, the experimental group will be counseled about their modified diet (very low carbohydrate diet <10%,40-50% protein and lipid in diet). Control group will be allowed to continue their routine diet counselled as part of their antenatal care.

ELIGIBILITY:
Inclusion Criteria:

* 2nd trimester women with GDM
* Either taking or not taking oral hypoglycemic agent or insulin

Exclusion Criteria:

* Previously known type 1 or type 2 Diabetic patients
* Age less than 18 and above 40 years
* Any other chronic disease

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Asses change in Fasting blood glucose | Baseline after one month and two month
Asses change in Postprandial glucose | Baseline after one month and two month
Asses change in Glycated hemoglobin A1c (HbA1c) | Baseline after one month and two month
Asses change in Lean and fat body mass | Baseline after one month and two month
Asses change in Fasting insulin | Baseline after one month and two month
Asses change in HOMA-IR | Baseline after one month and two month
Asses change in Adiponectin | Baseline after one month and two month
Carboxymethyl-lysine | Baseline after one month and two month
Asses change in C-reactive protein | Baseline after one month and two month
Asses change in NFk | Baseline after one month and two month

CONTACTS AND LOCATIONS:
Locations (1):
- Khyber Medical University, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Trout KK, Homko CJ, Wetzel-Effinger L, Mulla W, Mora R, McGrath J, Basel-Brown L, Arcamone A, Sami P, Makambi KH. Macronutrient Composition or Social Determinants? Impact on Infant Outcomes With Gestational Diabetes Mellitus. Diabetes Spectr. 2016 May;29(2):71-8. doi: 10.2337/diaspect.29.2.71. PMID 27182173
- [Background] Moreno-Castilla C, Hernandez M, Bergua M, Alvarez MC, Arce MA, Rodriguez K, Martinez-Alonso M, Iglesias M, Mateu M, Santos MD, Pacheco LR, Blasco Y, Martin E, Balsells N, Aranda N, Mauricio D. Low-carbohydrate diet for the treatment of gestational diabetes mellitus: a randomized controlled trial. Diabetes Care. 2013 Aug;36(8):2233-8. doi: 10.2337/dc12-2714. Epub 2013 Apr 5. PMID 23564917
- [Background] Mustad VA, Huynh DTT, Lopez-Pedrosa JM, Campoy C, Rueda R. The Role of Dietary Carbohydrates in Gestational Diabetes. Nutrients. 2020 Jan 31;12(2):385. doi: 10.3390/nu12020385. PMID 32024026
- [Background] Major CA, Henry MJ, De Veciana M, Morgan MA. The effects of carbohydrate restriction in patients with diet-controlled gestational diabetes. Obstet Gynecol. 1998 Apr;91(4):600-4. doi: 10.1016/s0029-7844(98)00003-9. PMID 9540949